CLINICAL TRIAL: NCT04979793
Title: Role of L-citrulline in Prevention of Pregnancy Associated Hypertension in Nulliparous Women
Brief Title: Role of L-citrulline in Prevention of Pregnancy Associated Hypertension
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: At the request of the PI
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-0167
Record Dates: First submitted 2021-06-16; First posted 2021-07-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Induced Hypertension; Preeclampsia and Eclampsia; Gestational Hypertension
Keywords: Pregnancy Induced Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Oral placebo, 3 grams milk powder sachet, taken once daily
  Interventions: Drug: Placebo
- Daily L-citrulline (Experimental): L-citrulline, 3 grams L-citrulline sachet, taken once daily
  Interventions: Drug: L-citrulline

INTERVENTIONS:
Drug: L-citrulline — 3 gram sachet, L-citrulline
  Arms: Daily L-citrulline
Drug: Placebo — Milk powder placebo
  Arms: Placebo

SUMMARY:
The target population for our study is healthy nulliparous pregnant women (first pregnancy) between the 12-16 week of pregnancy.

If a subject is eligible, written consent will be obtained by person to person contact. Eligible participants will be randomized to receive either daily L-citrulline supplementation or placebo.

DETAILED DESCRIPTION:
Healthy nulliparous pregnant women (first pregnancy) between the 12-16 week of pregnancy will be eligible for this study. The purpose of this study will be to determine if daily supplementation of oral L-citrulline can reduce the incidence of pregnancy induced hypertension. This will be a double blind study, subjects will be randomized to receive either L-citrulline (3 gram sachet) or a placebo for a total of 8 weeks. Participants will be asked to provide urine and blood samples at time of enrollment, be asked to respond to a phone survey to assess for side effects, and again be asked to provide urine and blood samples at the end of 8 weeks. Participants will continue with routine prenatal care throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous (no previous pregnancy greater than 20 weeks)
* Gestational age of pregnancy between 12 and 16 weeks

Exclusion Criteria:

* Known fetal anomaly or chromosomal abnormality
* Early fetal growth restriction
* Fetal demise or planned termination
* Participation in another study that may influence this study
* Known maternal kidney disease
* Known maternal electrolyte imbalance
* Known allergies to study interventions
* Preexisting hypertension (chronic hypertension)
* Known gastric ulcer
* Incarcerated status
* Planned delivery at non-UTMB hospital
* Known lactose intolerance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pregnancy induced hypertension | To be assessed by chart review at time of delivery which generally will occur 8-9 months after randomization.
  Incidence of pregnancy induced hypertension conditions (gestational hypertension, preeclampsia, or eclampsia) between treatment and placebo groups will be assessed by chart review after end of pregnancy

SECONDARY OUTCOMES:
Change in bioavailability of L-citrulline and asymmetric dimethyl arginine (ADMA) with oral L-citrulline administration | Baseline at start of study and again after 8 weeks treatment
  Assessment of change in serum L-citrulline and asymmetric dimethyl arginine (ADMA ) levels with L-citrulline administration between treatment and placebo groups. Serum samples will be collected at the beginning of study and after 8 weeks and assayed for ADMA and L-citrulline
Change in maternal nitric oxide levels with L-citrulline supplementation | Baseline at start of study and again after 8 weeks treatment
  Assessment of change in nitric oxide levels between treatment and placebo groups by measurement of baseline and 8 week post treatment urine nitrate and nitrite concentrations
Maternal blood pressure | Baseline at start of study, and approximately every 1-4 weeks after randomization at prenatal appointments throughout pregnancy. Also at time of delivery approximately 8-9 months after randomization..
  Assessment of maternal blood pressure throughout study
Maternal Morbidity | To be assessed by chart review at time of delivery which generally will occur 8-9 months after randomization.
  Composite assessment of incidence of maternal outcomes to include development of preeclampsia; Hemolysis, Elevated liver enzymes, Low Platelets (HELLP) syndrome; eclampsia; indicated preterm birth less than 32 weeks due to hypertension related disorders
Birth weight | To be assessed by chart review at time of delivery which generally will occur 8-9 months after randomization.
  To assess the actual birthweight of neonate by chart review at time of delivery. This outcome is different than fetal growth restriction noted in outcome 5.
Neonatal Outcomes | To be assessed by chart review 8-9 months after enrollment at time of delivery
  To determine the incidence of neonatal outcomes by chart review after delivery that include respiratory distress syndrome, necrotising enterocolitis, bronchopulmonary dysplasia (BPD), and BPD related pulmonary hypertension, retinopathy of prematurity, age at full feed, and length of hospital stay, fetal growth restriction defined as less than 10% of predicted gestational age, fetal death after 20 weeks gestation, and neonatal death

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No